CLINICAL TRIAL: NCT04643847
Title: Upfront Radiotherapy Combined With Almonertinib for Brain Metastasis in Non-small Cell Lung Cancer With EGFR Mutation: A Prospective Single-arm Phase II Trial
Brief Title: A Phase II Trial of Upfront Radiotherapy Plus Almonertinib for Epidermal Growth Factor Receptor(EGFR)-Mutant Non-small-cell Lung Cancer(NSCLC) Patients With Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AlmonRad
Record Dates: First submitted 2020-11-15; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: EGFR Positive Non-small Cell Lung Cancer; Brain Metastases
Keywords: NSCLC; EGFR; Brain metastasis
MeSH Terms: conditions — Brain Neoplasms | interventions — aumolertinib

STUDY DESIGN:
Intervention Model Description: 110mg Almonertinib is administered orally daily since the first day after stereotactic radiosurgery treatment (total dose 30 Gy, 5 fractions, day1, 3, 5, calibrated by cone beam computed tomography(CBCT) before each treatment). For patients who are assessed as oligometastasis three month after Almonertinib treatment, stereotactic body radiation therapy(SBRT) is recommended for oligometastatic lesions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic radiosurgery with Almonertinib (Experimental): 110mg Almonertinib is administered orally daily since the first day after stereotactic radiosurgery treatment (total dose 30 Gy, 5 fractions, day1, 3, 5, calibrated by CBCT before each treatment). For patients who are assessed as oligometastasis three months after Almonertinib treatment, SBRT is recommended for oligometastatic lesions
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — 110mg Almonertinib is administered orally daily since the first day after stereotactic radiosurgery treatment (total dose 30 Gy, 5 fractions, day1, 3, 5, calibrated by CBCT before each treatment). For patients who are assessed as oligometastasis three months after Almonertinib treatment, SBRT is recommended for oligometastatic lesions (The number of lesions received SBRT and radiation dose are not standardized).
  Other Names: HS-10296

SUMMARY:
Almonertinib is a three-generation epidermal growth factor receptor tyrosine kinase inhibitor(EGFR-TKI), which has shown competitive potential in the second-line treatment against first-generation TKIs. This study intends to assess the efficacy and safety of stereotactic radiosurgery with sequential almonertinib in treatment-naive EGFR-mutant NSCLC patients with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or pathologically confirmed non-small-cell lung cancer (adenocarcinoma).
2. The presence of radiographically definite brain metastases and intracranial foci measurable according to the RANO-BM criteria.
3. The number of brain metastases ≤ 10, the volume of individual metastases ≤ 15 cc, the diameter of individual metastases ≤ 30 mm, the diameter of metastases in the brainstem ≤ 5 mm, distance of the foci from the optic nerve, or optic cross > 5 mm.
4. EGFR-sensitive mutations (include 19del or L858R mutation or coexist with other types of EGFR mutation).
5. Comply with the indications and drug instructions for first-line treatment with a third-generation EGFR-TKI.
6. Have not received systemic antineoplastic therapy, excluding neoadjuvant, adjuvant, or synchronous chemotherapy more than 6 months prior to enrollment.
7. Asymptomatic or mildly symptomatic brain metastases (e.g., headache, nausea, or seizures for which dexamethasone/analgesic/antiepileptic medication is effective and sustained at a steady dose for 3 days or more).
8. Age ≥ 18 years.
9. Eastern Cooperative Oncology Group (ECOG) performance status(PS) score ≤ 2.
10. Survival is expected to be ≥ 6 months.
11. Women must use contraception after surgical sterilization, after sterilization, or during and for three months after treatment.
12. With informed consent signed.

Exclusion Criteria:

1. Previous treatment with almonertinib or other EGFR-TKI.
2. Patients with symptomatic brain metastases resulting in neurological deficits (not including headaches, nausea, or controlled seizures).
3. Multiple sclerosis.
4. Pacemakers implanted in the body or metals that cannot be examined by MRI.
5. Allergy to magnetic resonance contrast agents.
6. Brain metastases requiring surgical decompression.
7. Meningeal metastases.
8. Previous radiotherapy or surgery for brain metastases.
9. Contraindications to radiotherapy for uncontrolled systemic lupus erythematosus, scleroderma, or other connective tissue diseases.
10. Other malignant neoplasms (except non-melanoma skin cancer and cervical cancer) within five years.
11. Any medical or non-medical reason that prevents the patient from continuing to participate in research.
12. It is expected that the patient will not be able to comply with the procedures, restrictions, and requirements of the study and the investigator determines that the patient is unfit to participate in the study.
13. Received studying drugs within 5 half-lives or 3 months, whichever is greater.
14. Currently receiving drugs or herbal supplements known to be potent inducers of Cytochrome P450 3A4(CYP3A4) or unable to be discontinued prior to receiving the first dose of study treatment) (at least 3 weeks prior).
15. The patient is taking any drug known to prolong the QT interval and cannot be discontinued until treatment with amitriptyline.
16. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Central nerve system duration of response（CNS DOR） | 1 year
  Central nerve system duration of response assessed by RANO-BM criteria

SECONDARY OUTCOMES:
Intracranial prgression-free survival(PFS) | 1 year
  Intracranial progression free survival assessed by Response Assessment in Neuro-Oncology Brain Metastases(RANO-BM) criteria
Intracranial response rate(RR） | 1 year
  Intracranial response rate assessed by RANO-BM criteria
Extracranial RR | 1 year
  Extracranial response rate assessed by Response Evaluation Criteria in Solid Tumors(RECIST) criteria
overall survival (OS) | 1 year
  overall survival
Neurocognitive function assessed by mini-mental state examination(MMSE) questionnaire score | 1 year
  Neurocognitive function assessed by mini-mental state examination(MMSE) questionnaire score
quality of life(QoL) assessed by EORTC QLQ-C30 | 1 year
  Quality of Life assessed by The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire core 30(EORTC QLQ-C30)
quality of life(QoL) assessed by EORTC QLQ-BN20 | 1 year
  Quality of Life assessed by The European Organization for Reasearch and Treatment of Cancer Quality of Life Questionnaire Brain Cancer 20(BN20)

OTHER OUTCOMES:
Intracranial RR accessed by volumetric criteria | 1 year
  Intracranial response rate accessed by volumetric criteria
intracranial progression rate assessed by brain MRI at 1year | 1 year
  intracranial progression rate assessed by brain MRI at 1year

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No